CLINICAL TRIAL: NCT03541317
Title: Improving Student Mental Health: Adaptive School-based Implementation of CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Amy M. Kilbourne, Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R01MH11420301
Record Dates: First submitted 2018-05-17; First posted 2018-05-30 (Actual); Results first posted 2021-07-26 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Depression; Anxiety
Keywords: Adaptive implementation; Coaching; Facilitation; School mental health; Implementation intervention
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stage 1: Optimal First Line Implementation Strategy (Experimental): All schools enrolled will first be randomized to an optimal first line treatment in order to compare REP vs. REP + Coaching. Schools assigned to Stage 1 treatment "REP" will receive a daylong didactic training covering core elements of CBT and proper screening and identification of students; training to help SPs identify eligible students; a package that includes tools to deploy CBT; and ongoing technical assistance in CBT implementation. Schools assigned to Stage 1 treatment "REP + Coaching" will receive the REP components plus weekly visits from a CBT expert or "Coach", for a minimum of 12 weeks.
  Interventions: Behavioral: Stage 1 Strategy: REP; Behavioral: Stage 1 Strategy: REP + Coaching
- Stage 2: Added Value of Providing Facilitation (Experimental): After 2 months, schools will be assessed to determine whether they could benefit from augmenting their current strategy with a step-up strategy called "Facilitation". Schools identified as potentially benefiting will be re-randomized to compare the added value of augmenting their current strategy with Facilitation, compared to continuing with their same strategy. Stage 2 treatment strategy: step-up will include provision of an additional implementation strategy called "Facilitation". A full-time Facilitator who is a member of the study team and has expertise in CBT, implementation methods, and use of EBPs in schools will support school professionals in strategic thinking and leadership skills to address organizational barriers. Sites receiving Facilitation will receive regular calls for up to a minimum of 10 weeks from the Facilitator. All schools will also continue to receive their first line treatment (i.e. REP or REP + Coaching).
  Interventions: Behavioral: Stage 2 Strategy: Augment with Facilitation; Behavioral: Stage 2 Strategy: No augmentation

INTERVENTIONS:
Behavioral: Stage 1 Strategy: REP — Schools will receive a daylong didactic training covering core elements of CBT and proper screening and identification of students; training to help SPs identify eligible students; a package that includes tools to deploy CBT; and ongoing technical assistance in CBT implementation.
  Arms: Stage 1: Optimal First Line Implementation Strategy
Behavioral: Stage 1 Strategy: REP + Coaching — Schools will receive a daylong didactic training covering core elements of CBT and proper screening and identification of students; training to help SPs identify eligible students; a package that includes tools to deploy CBT; ongoing technical assistance in CBT implementation; and weekly visits from a CBT expert or "Coach", for a minimum of 12 weeks.
  Arms: Stage 1: Optimal First Line Implementation Strategy
Behavioral: Stage 2 Strategy: Augment with Facilitation — In addition to first-line treatment (REP or REP + Coaching), schools will also receive support from a Facilitator who is a member of the study team and has expertise in CBT, implementation methods, and use of EBPs in schools will support SPs in strategic thinking and leadership skills to address organizational barriers.
  Arms: Stage 2: Added Value of Providing Facilitation
Behavioral: Stage 2 Strategy: No augmentation — Schools will continue to receive their first-line treatment (REP or REP + Coaching); no additional support will be offered.
  Arms: Stage 2: Added Value of Providing Facilitation

SUMMARY:
The overarching goal of this study is to improve the delivery of an established, evidence-based intervention (cognitive-behavioral therapy-CBT) in Michigan schools through different implementation strategies designed to better educate school professionals. Specifically, the study will assist the ongoing Transforming Research into Action to Improve the Lives of Students (TRAILS) Program by evaluating different ways to educate school professionals (SPs) to improve their delivery of CBT to high school students and ultimately improve student mental health outcomes in the state of Michigan. The three educational approaches are Replicating Effective Programs (REP), Coaching, and Facilitation.

DETAILED DESCRIPTION:
This study seeks to develop an effective and efficient sequence of implementation strategies for encouraging delivery of Cognitive Behavioral Therapy (CBT) by school professionals in high schools across Michigan. In the run-in phase, all schools will receive support and training from REP for three months. After three months, schools will be randomized to either (1) continue with REP; or (1) augment REP with a minimum of 12 weeks of coaching. Eight weeks after this first randomization, schools will be evaluated to determine whether they might also benefit from an augmentation of their current strategy with Facilitation. Schools that could benefit from Facilitation (defined as delivering 3 or more CBT modules to less than 10 students or reporting 3 or more organizational barriers to delivering CBT) will be re-randomized to either (1) continue with their current strategy (REP or REP + Coaching); or (2) have their current strategy augmented with Facilitation. All implementation support will be discontinued 12 months after first randomization; outcomes will be assessed through 18 months after study start.

This results in four sequences of implementation strategies: REP only; REP + Facilitation for those who did not adequately respond initially to REP alone; REP + Coaching; and REP + Coaching + Facilitation for those who did not adequately respond initially to REP + Coaching.

ELIGIBILITY:
School Administrators

Inclusion Criteria:

* Working at a school that is located within a 2-hour drive of a TRAILS coach
* Employed at a Michigan high school full or part time
* Able to read and understand English

Exclusion Criteria:

* Unable to provide informed consent for participation in the study activities

School Professional

Inclusion Criteria:

* Working at a school that is located within a 2-hour drive of a TRAILS coach
* Employed at a Michigan high school full or part time
* Have a background in clinical school social work, counseling, psychology, or similar area
* Able to read and understand English

Exclusion Criteria:

* Has previously received coaching in CBT through the TRAILS or similar programs
* Has a significant illness or condition that precludes their participation in the implementation strategies, including the REP training and student identification process, Coaching, or Facilitation
* Unable to provide informed consent for participation in the study activities

Student

Inclusion Criteria:

* Age 14-21 years
* Currently enrolled in the 9th, 10th, or 11th grade at time of first assessment at one of the participating schools
* Have at least one symptom of depression or anxiety that impacts their daily well-being or functioning, as determined by the SP
* Able to read and understand English and comprehend assessments

Exclusion Criteria:

* Evidence of psychosis, as identified by any standardized measure; reported by the student, parent, or referral source; or noted by the SP during the recruitment and screening process
* Evidence of a severe pervasive developmental disability, mental retardation or other cognitive impairment that would interfere with the potential for benefit from skills groups, as identified by the student, parent, or referral source.
* Unable to attend CBT group sessions

Students could withdraw from participation at any time by themselves, or by parent notification to the study team.

Ages: 14 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1329 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy M Kilbourne, PhD, MPH, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Smith SN, Almirall D, Choi SY, Andrews C, Koschmann E, Rusch A, Bilek EL, Lane A, Abelson JL, Eisenberg D, Himle JA, Liebrecht C, Kilbourne AM. Student mental health outcomes of a clustered SMART for developing an adaptive implementation strategy to support school-based CBT delivery. J Affect Disord. 2024 Dec 15;367:399-407. doi: 10.1016/j.jad.2024.08.048. Epub 2024 Aug 14. PMID 39151756
- [Derived] Smith SN, Almirall D, Choi SY, Koschmann E, Rusch A, Bilek E, Lane A, Abelson JL, Eisenberg D, Himle JA, Fitzgerald KD, Liebrecht C, Kilbourne AM. Primary aim results of a clustered SMART for developing a school-level, adaptive implementation strategy to support CBT delivery at high schools in Michigan. Implement Sci. 2022 Jul 8;17(1):42. doi: 10.1186/s13012-022-01211-w. PMID 35804370
- [Derived] Kilbourne AM, Smith SN, Choi SY, Koschmann E, Liebrecht C, Rusch A, Abelson JL, Eisenberg D, Himle JA, Fitzgerald K, Almirall D. Adaptive School-based Implementation of CBT (ASIC): clustered-SMART for building an optimized adaptive implementation intervention to improve uptake of mental health interventions in schools. Implement Sci. 2018 Sep 5;13(1):119. doi: 10.1186/s13012-018-0808-8. PMID 30185192

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 1329 consented, listed in registration: there were 103 School administrators (for 94 schools), 978 Students were enrolled into the study, 227 school professionals from 115 schools were enrolled/consented; 21 coaches were also consented.
  Because primary and secondary outcome measures are all based on data collected from school professionals, only they are included in participant flow, baseline characteristics, outcome measures.
Pre-assignment Details: Pre-randomization, 21 schools and a total of 58 school professionals declined or did not meet eligibility and were dropped.
  Stage 1 Randomization: 94 schools (employing 169 school professionals (SPs)) were enrolled in the sequentially-randomized trial.
  Stage 2 Randomization: All 83 schools (employing 154 SPs) identified as potentially benefitting from augmentation with Facilitation (i.e., "schools that did not respond sufficiently following Stage 1 strategy") were re-randomized at Stage 2.
Units Other Than Participants: Schools
Groups:
- REP Only, Responders, Continue: This group included schools who responded sufficiently to "REP only" in Stage 1, and then were assigned to Continue "REP only" in Stage 2.
- REP Only, Non-responders, Continue: This group included schools who did not respond sufficiently to "REP only" in Stage 1, and then were assigned to Continue "REP only" in Stage 2.
- REP Only, Non-responders, Facilitation: This group included schools who did not respond sufficiently to "REP only" in Stage 1, and then were assigned to Augment "REP" with "Facilitation" in Stage 2.
- REP + Coaching, Responders, Continue: This group included schools who responded sufficiently to "REP + Coaching" in Stage 1, and then were assigned to Continue "REP + Coaching" in Stage 2.
- REP + Coaching, Non-responders, Continue: This group included schools who did not respond sufficiently to "REP + Coaching" in Stage 1, and then were assigned to Continue "REP + Coaching" in Stage 2.
- REP + Coaching, Non-responders, Facilitation: This group included schools who did not respond sufficiently to "REP + Coaching" in Stage 1, and then were assigned to Augment "REP + Coaching" with "Facilitation" in Stage 2.
Period: Stage 1 of the Implementation
Arm/Group | REP Only, Responders, Continue | REP Only, Non-responders, Continue | REP Only, Non-responders, Facilitation | REP + Coaching, Responders, Continue | REP + Coaching, Non-responders, Continue | REP + Coaching, Non-responders, Facilitation
Started | 6; 5 Schools | 37; 21 Schools | 38; 21 Schools | 9; 6 Schools | 43; 21 Schools | 36; 20 Schools
Completed | 6; 5 Schools | 37; 21 Schools | 38; 21 Schools | 9; 6 Schools | 43; 21 Schools | 36; 20 Schools
Not Completed | 0; 0 Schools | 0; 0 Schools | 0; 0 Schools | 0; 0 Schools | 0; 0 Schools | 0; 0 Schools
Period: Stage 2 of the Implementation
Arm/Group | REP Only, Responders, Continue | REP Only, Non-responders, Continue | REP Only, Non-responders, Facilitation | REP + Coaching, Responders, Continue | REP + Coaching, Non-responders, Continue | REP + Coaching, Non-responders, Facilitation
Started | 6; 5 Schools | 37; 21 Schools | 38; 21 Schools | 9; 6 Schools | 43; 21 Schools | 36; 20 Schools
Completed | 5; 5 Schools | 37; 21 Schools | 38; 21 Schools | 9; 6 Schools | 43; 21 Schools | 36; 20 Schools
Not Completed | 1; 0 Schools | 0; 0 Schools | 0; 0 Schools | 0; 0 Schools | 0; 0 Schools | 0; 0 Schools
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Demographic data is presented for school professionals when human data is needed, because that is the group on which all primary and secondary outcome measures are based. Some baseline characteristics apply to school units rather than to school professionals.
Units Other Than Participants: schools
Groups:
- Stage 1 Strategy: REP:: Stage 1 Strategy: REP. This includes all three arms listed in Participant Flow as not receiving Coaching
- Stage 1 Strategy: REP + Coaching: Stage 1 Strategy: REP + Coaching This includes all three arms listed in Participant Flow as receiving Coaching.
- Total: Total of all reporting groups
Arm/Group | Stage 1 Strategy: REP: | Stage 1 Strategy: REP + Coaching | Total
Number analyzed (Participants) | 81 | 88 | 169
Number analyzed (schools) | 47 | 47 | 94
Age, Customized [Count of Participants; unit: Participants] — Age data was not collected from School Professionals, but all had to be adults to be in their roles.
  Participants
    > 18 years of age | 81 | 88 | 169
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 69 | 74 | 143
  Male | 8 | 12 | 20
  Unknown | 4 | 2 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white | 71 | 80 | 151
  non-white | 5 | 6 | 11
  unknown | 5 | 2 | 7
Rural schools (vs urban) (Binary proportion) [Mean (Standard Deviation); unit: proportion] — rural (1) or urban (0) Population: This baseline characteristic applies to school units rather than to school professionals. All participating schools are included in the analysis.
  proportion
    number analyzed (Participants) | 47 | 47 | 94
    (all) | .55 (.50) | .57 (.50) | .56 (.50)
Schools with > 500 students (vs. ≤ 500 students), Binary Proportion [Mean (Standard Deviation); unit: proportion] — > 500 students (1) or ≤ 500 students (0) Population: As this baseline characteristic applies to schools, not to the school professionals who participated in the study, number of schools analyzed is shown. All schools are included.
  proportion
    number analyzed (Participants) | 47 | 47 | 94
    (all) | 0.66 (0.48) | 0.64 (0.49) | 0.65 (0.48)
Schools with ≥ 50% of students on free/reduced cost lunch [Mean (Standard Deviation); unit: proportion] — ≥ %50 (1) or < 50% (0), Binary proportion
  proportion | 0.36 (0.49) | .36 (.49) | .36 (.48)
School level average School Professional tenure [Mean (Standard Deviation); unit: years] | 7.34 (6.03) | 7.79 (5.94) | 7.56 (5.96)
School level Proportion of School Professionals with graduate degree [Mean (Standard Deviation); unit: Proportion] | .89 (.28) | .91 (.24) | .90 (.26)

OUTCOME MEASURES:

1. Primary Outcome: Number of CBT Sessions Delivered by School Professionals to Students After 18 Months
Description: School professionals include counselors, social workers, and trained mental health providers working within the school. The primary aim is a comparison of schools offered the REP only intervention (the least intensive strategy) versus schools offered the adaptive implementation strategy involving REP, Coaching, and Facilitation (the most intensive strategy).
Time Frame: Baseline to 18-months
Population: The primary outcome measure pertains to delivery of CBT by school professionals only, and thus the number analyzed reflects data categorized by number of school professionals that had REP only vs. most intensive intervention: REP, Coaching and Facilitation
Measure: Mean (95% Confidence Interval); unit: number of CBT sessions
Units Other Than Participants: schools
Groups:
- Group 1: REP Only: This arm consists of only those professionals in schools that received REP only: including those who were originally randomized to receive REP only and never re-randomized to receive facilitation ("responders" to REP) and those who were "non-responders to REP" but randomized to continue with REP only in Stage 2. Thus, it corresponds in Participant Flow to both the REP only, Responders Continue and REP Only, Non-Responders Continue. The 43 professionals represent 26 schools.
- Group 2: REP + Coaching, Responders Continue and REP + Coaching With Facilitation: This arm consists of those schools that received REP + Coaching in Stage 1, who were either Responders after Stage 1 or, as Non-Responders were randomized to additionally receive "Facilitation" in Stage 2. A full-time Facilitator who is a member of the study team and has expertise in CBT, implementation methods, and use of EBPs in schools supported school professionals in strategic thinking and leadership skills to address organizational barriers. Sites receiving Facilitation received regular calls for a minimum of 10 weeks from the Facilitator.
  Thus, this arm represents "REP + Coaching Responders, Continue" and "REP + Coaching, Non-Responders, Facilitation" from the Participant Flow. The 45 professionals represent 26 schools.
Arm/Group | Group 1: REP Only | Group 2: REP + Coaching, Responders Continue and REP + Coaching With Facilitation
Number analyzed (Participants) | 43 | 45
Number analyzed (schools) | 26 | 26
number of CBT sessions | 121.1 [87.52 to 154.65] | 111.4 [86.63 to 136.16]
Statistical Analysis 1: Comparison: Group 1: REP Only vs Group 2: REP + Coaching, Responders Continue and REP + Coaching With Facilitation; Test type: Superiority — A test of the null hypothesis that there is no difference between these two strategies on the sum of the average number of CBT sessions delivered to students by SPs over the four post-randomization phases during Stages 1 and 2; p = 0.63, weighted least squares regression; Marginal means under each implementation strategy estimated after each of 4 post-randomization phases (NeCamp, Kilbourne, & Almirall 2017); Difference in sum of means* = 9.7, 95% CI 2-sided [-30.03 to 49.40] — *Difference in the sum of the means estimated at each post-randomization phase

2. Secondary Outcome: Number of Brief Individual CBT Sessions
Description: The sum of the average number of brief individual CBT sessions (<15 min.) delivered to students by SPs over all four post-randomization phases occurring during Stages 1 and 2.
Time Frame: 18 months
Measure: Mean (95% Confidence Interval); unit: Number of brief sessions
Units Other Than Participants: schools
Arm/Group | Group 1: REP Only | Group 2: REP + Coaching, Responders Continue and REP + Coaching With Facilitation
Number analyzed (Participants) | 43 | 45
Number analyzed (schools) | 26 | 26
Number of brief sessions | 55.9 [39.58 to 72.21] | 52.1 [38.56 to 65.67]
Statistical Analysis 1: Comparison: Group 1: REP Only vs Group 2: REP + Coaching, Responders Continue and REP + Coaching With Facilitation; Test type: Superiority — A test of the null hypothesis that there is no difference between these two strategies on the sum of the average number of brief individual CBT sessions (<15 min.) delivered to students by SPs over the four post-randomization phases occurring during Stages 1 and 2; p = 0.72, weighted least squares regression; Marginal means under each embedded implementation strategy estimated after each of 4 post-randomization phases (NeCamp, Kilbourne & Almirall 2017); Difference in sum of means* = 3.78, 95% CI 2-sided [-16.88 to 24.44] — *Difference in the sum of the means estimated at each post-randomization phase

3. Secondary Outcome: Number of Full Individual CBT Sessions
Description: The sum of the average number of full individual CBT sessions (≥15 min.) delivered to students by SPs over all four post-randomization phases occurring during Stages 1 and 2.
Time Frame: 18 Months
Measure: Mean (95% Confidence Interval); unit: full sessions
Units Other Than Participants: schools
Groups:
- Group 2: REP + Coaching, Responders Continue and REP + Coaching With Facilitation: This arm consists of those schools that received REP + Coaching in Stage 1, who were either Responders after Stage 1 or, as Non-Responders were randomized to additionally receive "Facilitation" in Stage 2. A full-time Facilitator who is a member of the study team and has expertise in CBT, implementation methods, and use of EBPs in schools supported school professionals in strategic thinking and leadership skills to address organizational barriers. Sites receiving Facilitation received regular calls for a minimum of 10 weeks from the Facilitator.
  Thus, this arm represents "REP + Coaching Responders" and "REP + Coaching with Facilitation" from the Participant Flow. The 45 professionals represent 26 schools.
Arm/Group | Group 1: REP Only | Group 2: REP + Coaching, Responders Continue and REP + Coaching With Facilitation
Number analyzed (Participants) | 43 | 45
Number analyzed (schools) | 26 | 26
full sessions | 49.5 [32.77 to 66.23] | 41.7 [29.07 to 54.23]
Statistical Analysis 1: Comparison: Group 1: REP Only vs Group 2: REP + Coaching, Responders Continue and REP + Coaching With Facilitation; Test type: Superiority — A test of the null hypothesis that there is no difference between these two strategies on the sum of the average number of brief individual CBT sessions (>15 min.) delivered to students by SPs over the four post-randomization phases occurring during Stages 1 and 2; p = 0.46, Weighted Least Squares Regression; [statistical method as in outcome 2, analysis 1]; Difference in sum of means* = 7.85, 95% CI 2-sided [-13.20 to 28.91] — Difference in the sum of the means estimated at each post-randomization phase

4. Secondary Outcome: Number of Group CBT Sessions
Description: The sum of the average number of group CBT sessions delivered to students by SPs over all four post-randomization phases occurring during Stages 1 and 2.
Time Frame: 18 Months
Measure: Mean (95% Confidence Interval); unit: group sessions
Units Other Than Participants: schools
Arm/Group | Group 1: REP Only | Group 2: REP + Coaching, Responders Continue and REP + Coaching With Facilitation
Number analyzed (Participants) | 43 | 45
Number analyzed (schools) | 26 | 26
group sessions | 16.8 [9.46 to 24.16] | 17.5 [14.03 to 20.92]
Statistical Analysis 1: Comparison: Group 1: REP Only vs Group 2: REP + Coaching, Responders Continue and REP + Coaching With Facilitation; A test of the null hypothesis that there is no difference between these two strategies on the sum of the average number of group CBT sessions delivered to students by SPs over the four post-randomization phase occurring during Stages 1 and 2; Test type: Superiority; p = 0.87, Weighted Least Squares Regression; [statistical method as in outcome 2, analysis 1]; Difference in sum of means* = -0.66, 95% CI 2-sided [-8.49 to 7.16] — Difference in the sum of the means estimated at each post-randomization phase

ADVERSE EVENTS:
Time Frame: 18 months
Description: AE Data was not collected for any group. While there was no request for school professionals to notify the study team about student adverse events, one professional spontaneously informed the team that one student had committed suicide from the REP Non-Responder, Facilitation group.
Groups:
- REP Only, Non-Responders, Continue: This group included schools who did not respond sufficiently to "REP only" in Stage 1, and were assigned to continue "REP only" in Stage 2.
- REP + Coaching Responders, Continue: This group included schools who responded sufficiently to "REP + Coaching" in Stage 1 and were assigned to continue "REP + Coaching" in Stage 2.
- REP+ Coaching Non-Responders, Continue: This group included schools who did not respond sufficiently to "REP + Coaching" in Stage 1 and were assigned to continue "REP + Coaching" in Stage 2.
- REP + Coaching, Non-Responders, Facilitation: This group included schools who did not respond sufficiently to "REP + Coaching" in Stage 1, and then were assigned to augment "REP+ Coaching" with "Facilitation" in Stage 2.
Arm/Group | REP Only, Responders, Continue | REP Only, Non-Responders, Continue | REP Only, Non-Responders, Facilitation | REP + Coaching Responders, Continue | REP+ Coaching Non-Responders, Continue | REP + Coaching, Non-Responders, Facilitation
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT03541317/Prot_SAP_000.pdf